CLINICAL TRIAL: NCT02357251
Title: Enhanced Recovery After Surgery: A Randomized Control Trial of Perioperative Management of Gynecologic Patients
Brief Title: Enhanced Recovery After Surgery: A RCT of Perioperative Management of Gynecologic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CASE 17814
Record Dates: First submitted 2015-02-03; First posted 2015-02-06 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Laparotomy; Gynecologic Diseases
MeSH Terms: conditions — Genital Diseases, Female

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced recovery protocol (Active Comparator): Aspects of perioperative care will be standardized. Specific protocol for pre-operative, intra-operative, and post-operative care will be followed in this group.
  Interventions: Other: Enhanced recovery protocol
- Standard of care (No Intervention): Treating physicians will determine all aspects of patients' perioperative care. Specifically, the individual surgeon, nurse, resident, fellow, and anesthesiologist caring for the patient will determine the patients' pre-operative counseling, bowel preparation, postoperative nausea and vomiting prophylaxis, IV fluid replacement, use of drains, timing of urinary catheter removal, mobilization, post-operative nutrition, pain medication, and bowel stimulation.

INTERVENTIONS:
Other: Enhanced recovery protocol
  Arms: Enhanced recovery protocol

SUMMARY:
This is a single-blinded randomized control trial comparing the current perioperative care of the investigators gynecologic oncology patients with a standardized perioperative "enhanced recovery" pathway. Adult patients undergoing laparotomy by one of the gynecologic oncology surgeons will be eligible to participate. The primary outcome will be length of hospitalization including any days of readmission in the 30 days post-operatively. Secondary outcomes will include 30-day readmission rate, complications, quality of recovery, and pain control.

DETAILED DESCRIPTION:
The objective of this research is to implement and evaluate an enhanced recovery pathway for gynecologic surgery patients undergoing laparotomy and compare their outcomes to the current standard of care perioperative management.

Hypothesis: Patients having a laparotomy for gynecologic disease have a shortened length of hospitalization in the 30 days post-operatively when undergoing a perioperative enhanced recovery protocol compared to the standard of care.

This study will be a randomized single-blinded control trial.

Primary Outcomes: Hospital days in first 30 days post-operatively (Length of stay of primary hospitalization plus any days of readmission)

Secondary Outcomes:

1. 30-day readmission rate
2. Complications as assessed by the incidence of a composite of major complications and a second composite of minor complications.
3. Patient reported quality of recovery and quality of life as determined by QoR-40 score and RAND-36 score.
4. Pain control at assessed by daily mean pain scores (scale 0-10) as elicited and recorded by nursing.

All women who meet inclusion criteria will be approached in the gynecologic oncology clinic at the completion of their appointment. Eligible patients that agree to participate will be provided written informed consent. The informed consent process will occur in a clinic exam room. There will be no other recruitment methods or advertisements employed. Patients can agree to participate at this time or at any time prior to their pre-operative teaching appointment which is scheduled at some point between their initial surgical consult visit and their surgery. The first study intervention will take place at their pre-operative teaching appointment and so enrollment must occur prior to this time.

Randomization will occur at study entry. The participants will then be randomized to one of two groups: "standard care" or "enhanced recovery care." Randomization will be stratified by disease type, age, and BMI. Given the longer length of hospitalization inherent in ovarian/primary peritoneal cancer debulking surgery, the investigators want to stratify based on the pre-operative suspected diagnosis in an attempt to balance these patients between groups. Similarly, advanced age and increased BMI are risks factors for peri-operative complications and increased length of hospitalizations and should be stratified between groups. Within each stratum, randomization will be performed in blocks of 8 to ensure that groups are balanced throughout the study in case recruitment goals are not reached. Two hundred randomization assignments will be assigned to each stratum to ensure sufficient assignments are available to each group in the event that more patients are recruited than expected.

Allocation will be revealed to the PI and the surgical team at the time of randomization. This is necessary because the pre-operative counseling intervention for those patients in the "enhanced recovery" intervention will need to occur at this time. Allocation will remain concealed for the patient and for the members of the research team who are conducting the post-discharge surveys.

Two survey instruments will be used to evaluate pre-operative and post-operative quality of life as well as quality of recovery. The RAND-36 will be utilized as a pre-operative and 4 week post-operative assessment of health-related quality of life. This 36 item health-related quality of life instrument includes eight dimensions: general health, physical functioning, emotional wellbeing, social functioning, energy, pain, and physical and emotional role functioning. While this is a generic assessment of quality of life and not designed to be specific to surgical recovery-related quality of life, the investigators are including this instrument in order to have a baseline health-related quality of life assessment of the investigators patients and to allow for comparisons to other studies of perioperative gynecology patients.

The QoR-40 is a 40-question tool used to evaluate the quality of recovery. It incorporates 5 dimensions of health: patient support, comfort, emotions, physical independence, and pain. The QoR40 is one of the most widely used measurements of patient-determined quality of recovery. It has been extensively validated and has excellent reliability, responsiveness, and clinical utility to a range of surgical settings.

Both the RAND-36 and QoR-40 have been used to study post-operative recovery in women undergoing gynecologic surgery and have been found to be valid. Furthermore, both surveys have been validated for both self-administration and telephone administration.

Description of Intervention Start of Study Interventions At their pre-operative teaching appointment, all study participants will be asked to complete a health and quality of life survey.

Protocol-specific Interventions:

1. "Standard of care" group: Treating physicians will determine all aspects of patients' perioperative care. Specifically, the individual surgeon, nurse, resident, fellow, and anesthesiologist caring for the patient will determine the patients' pre-operative counseling, bowel preparation, postoperative nausea and vomiting prophylaxis, IV fluid replacement, use of drains, timing of urinary catheter removal, mobilization, post-operative nutrition, pain medication, and bowel stimulation.
2. "Enhanced recovery" group: Aspects of perioperative care will be standardized in terms of the pre-operative, intra-operative and post-operative management of issues such as pre-operative counseling, bowel preparation, postoperative nausea and vomiting prophylaxis, IV fluid replacement, use of drains, timing of urinary catheter removal, mobilization, post-operative nutrition, pain medication, and bowel stimulation. Of note, these interventions have previously been studied in isolation and in combination. They are considered by many to be the standard perioperative management of surgical patients

Postoperative Interventions All participants will be surveyed post-surgery regarding their quality of recovery.

Post-discharge and Over-the-Phone Interventions Participants will be called 4 weeks after their surgery and asked about any hospital readmissions and complications at this time. They will also complete post-discharge surveys.

ELIGIBILITY:
Inclusion Criteria:

* patients who are to undergo laparotomy

Exclusion Criteria:

* Inability to provide informed consent
* Inability to comprehend written or spoken English
* Immobility as defined by inability to ambulate unassisted
* Patient currently residing in a skilled nursing facility
* ASA physical status 4 or 5
* Planned greater than one night admission to the ICU
* Pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-12-12 (Actual); Primary Completion 2017-07-03 (Actual); Study Completion 2017-07-03 (Actual)

PRIMARY OUTCOMES:
Length of hospitalization | 30 days post-operatively
  Hospital days in first 30 days post-operatively (Length of stay of primary hospitalization plus any days of readmission)

SECONDARY OUTCOMES:
Readmission rate | 30 days post-operatively
Complications | 30 days post-operatively
  as assessed by the incidence of a composite of major complications and a second composite of minor complications.
  Major complications: Deep surgical site infection, Organ/space infection, Sepsis, Bowel perforation, obstruction and/or anastomotic leak, Bleeding, Internal or external fistula formation, Pulmonary emboli (PE), Pulmonary edema with congestive heart failure, Acute heart failure, Myocardial infarction, Ventricular arrhythmias, Renal failure, Respiratory failure (including aspiration), Pneumonia
  Minor complications: Superficial incisional surgical site infection, Postoperative fever, Unplanned ICU admission, Non-ventricular arrhythmias, Paralytic Ileus, DVT, Cystitis or urinary tract infection, Urinary retention, Hemodynamic disturbances, Renal insufficiency, Transient neurological complication
Quality of life/recovery | 30 days post-operatively
  Patient reported quality of recovery and quality of life as determined by QoR-40 score and RAND-36 score
Pain control | 30 days post-operatively
  Pain control at assessed by daily mean pain scores (scale 0-10) as elicited and recorded by nursing.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Maurer, MD, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States